CLINICAL TRIAL: NCT03658070
Title: A Phase I Open and Multiple Ascending Dose Study to Assess the Safety、Tolerability、Pharmacokinetics and Pharmacodynamic Characteristics of XY0206 in Subjects With Chinese Advanced or Metastatic Solid Tumours
Brief Title: A Study of XY0206 in Subjects With Advanced or Metastatic Solid Tumours
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shijiazhuang Yiling Pharmaceutical Co. Ltd (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XY0206ONC1001
Record Dates: First submitted 2018-08-08; First posted 2018-09-05 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Advanced or Metastatic Solid Tumours

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- XY0206-12.5mg (Experimental): Drug:XY0206;Dosage form:Tablet;Dosage：12.5mg;Include single dose treatment and multiple dose phase
  Interventions: Drug: XY0206
- XY0206-25mg (Experimental): Drug:XY0206;Dosage form:Tablet;Dosage：25mg;Include single dose treatment and multiple dose phase
  Interventions: Drug: XY0206
- XY0206-37.5mg (Experimental): Drug:XY0206;Dosage form:Tablet;Dosage：37.5mg;Include single dose treatment and multiple dose phase
  Interventions: Drug: XY0206
- XY0206-50mg (Experimental): Drug:XY0206;Dosage form:Tablet;Dosage：50mg;Include single dose treatment and multiple dose phase
  Interventions: Drug: XY0206
- XY0206-75mg (Experimental): Drug:XY0206;Dosage form:Tablet;Dosage：75mg;Include single dose treatment and multiple dose phase
  Interventions: Drug: XY0206
- XY0206-100mg (Experimental): Drug:XY0206;Dosage form:Tablet;Dosage：100mg;Include single dose treatment and multiple dose phase
  Interventions: Drug: XY0206

INTERVENTIONS:
Drug: XY0206 — Dosage form:Tablet;Single dose treatment:Take the drug once on day 1,each time 1 tablet. Multiple dose phase:Take the medicine once a day,1 tablet at a time.4 weeks of continuous medication is one course of treatment. After the first course of treatment, the subjects can continue to receive the experimental drug treatment until they meet the criteria for stopping treatment or determine the duration and interval of treatment according to the accumulated condition after multiple dose.

SUMMARY:
1. To observe the safety and tolerability of oral XY0206 in patients with advanced/metastatic malignant solid tumor in China, and observe the drug dose limiting toxicity (DLT) to establish the maximum tolerated dose (MTD) in humans.
2. To investigate the pharmacokinetic (PK) characteristics, pharmacodynamics (PD) characteristics, and PK/PD correlation of single and multiple doses of XY0206 in patients with advanced/metastatic malignant solid tumors to provide dose selection basis for clinical studies;
3. To evaluate the effect of standard meal on main PK parameters of XY0206;
4. To determine the metabolites of XY0206 in patients with advanced/metastatic malignant solid tumor.
5. To explore the correlation between PK and QTcF.
6. Preliminary investigates the effectiveness of XY0206 in patients with advanced/metastatic malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria before entering the group:

  1. Patients with advanced/metastatic solid tumor (such as non-small cell lung cancer, gastrointestinal stromal tumor, renal cell carcinoma, pancreatic cancer, etc.) who have failed standard treatment with histological or cytological diagnosis, have no effective treatment, or have relapsed after treatment.
  2. Patients with measurable or evaluable tumor lesions (1.1 version of RECIST efficacy evaluation criteria).
  3. The age is 18~70 years old (including upper and lower limit), and there is no restriction on male and female (for participating in the extended trial)Of patients with a sex ratio of not less than 30%).
  4. Physical condition ECOG≤2.
  5. Expected survival ≥3 months.
  6. BMI at 19≤BMI≤30, BMI = weight (kg)/height 2 (m2).
  7. Liver function: AST <2.5×ULN, ALT<2.5×ULN, total bilirubin <1.5×ULN.
  8. Blood biochemistry: Serum potassium and sodium levels are within the range of normal laboratory values (if researchers and physiciansThe overseer assesses results beyond the normal range to be of no clinical significance and the patient canInto the group; If the drug can be controlled within the normal range during the screening period, the patient canTo enroll).
  9. Renal function: serum creatinine (Scr) ≤1.5×ULN or calculated creatinine clearance rate(Ccr) >60mL/min Ccr calculation formula: male Ccr=[(140- age)× weight(kg)] / [0.818 x Scr (mu mol/L)], women Ccr = 0.85 x [(140 - age) by weight(kg)] / [0.818 x Scr (mu mol/L)].
  10. blood routine: platelet count of > 80×109/L, hemoglobin of > 90g/L, neutrophil pair count of > 1.5×109 /L.
  11. Urine routine: urinary protein - or 1+, or 24-hour urinary protein <1 g [Note: if due to urinary tractTransient abnormalities of the above urinary protein due to infection and other causes returned to normal after retesting.You can also consider enrolling; Subjects without proteinuria symptoms may also be considered for inclusion.
  12. Coagulation function: International standardized ratio < 1.5.
  13. No other antitumor concomitant therapy (including steroids with antitumor effects).
  14. Women of childbearing age and men agreed to use it throughout the study period and within 6 months after completion of treatmentRegular contraception that is effective enough.
  15. Understand and voluntarily sign written informed consent, and have the willingness and ability to complete regular visits and treatmentTreatment planning, laboratory examination and other test procedures.

Exclusion Criteria:

* Patients cannot participate in this clinical study if they meet any of the following conditions:

  1. Pregnant or lactating women.
  2. Tested positive for human immunodeficiency virus (HIV).
  3. The active period of HBV or HCV infection is known to be associated with abnormal liver function, and antiviral drugs are required.
  4. Severe trauma, ulcer or fracture at screening time.
  5. A history of uncontrolled epilepsy, central nervous system disease or mental illness.
  6. Symptomatic or uncontrolled brain metastases or meningeal diseases.
  7. diabetes or hypertension with poor drug control (under optimal drug treatment, fasting blood glucose >7mmol/L, or blood pressure > 150/100mmhg).
  8. Uncontrolled thyroid dysfunction.
  9. Persistent arrhythmias of version 4.03 or above, NCI CTCAE level ≥2, atrial fibrillation of any level.
  10. Cardiac ejection fraction (ECHOcardiography) below 50%.
  11. patients with clinically significant prolonged history of QTc (>450ms for male and >470ms for female).
  12. Have a history of severe drug allergy (NCI CTCAE level ≥3 according to version 4.03 or above) and may be allergic to test drug ingredients; Has been treated with or is allergic to sunitinib malate.
  13. for the first time to give medicine taken within 4 weeks before have significant effects on P450 metabolic pathway of drugs (for example: ketoconazole, itraconazole, clarithromycin, aza that wei, indiana that wei, naphthalene sanzuotong, that of the wei and the wey, ShaKui the wey, terry toxin, voriconazole, dexamethasone, phenytoin, carbamazepine, rifampicin, dean, rifampicin and dean at the cloth, phenobarbital, st. John's wort, etc.) or to eat within 48 h before delivery of P450 metabolic enzyme pathways have a significant impact on food (such as grapefruit and food containing grapefruit).
  14. Received any experimental drug therapy within 6 weeks prior to initial administration.
  15. for the first time six weeks before the treatment, patients treated with anti-tumor therapy (chemotherapy, radiation therapy, biological therapy, or hormone therapy) (note: for anti-tumor small molecules targeting drugs, if the patient before the first test drugs, always use small molecules targeting drug has cleared more than 5 half-life, the patient may also be considered into the group]. Surgery was performed within 14 weeks prior to the first administration.
  16. patients have any limit test compliance of medical or psychiatric conditions, such as the central nervous system (CNS) leukemia, active control of bacterial infection, 3, or 4 bleeding, unstable angina, myocardial infarction, stroke or transient ischemic attack, pulmonary embolism, or into the group of six months before the test of catheter-related deep vein thrombosis, insulin-dependent diabetes mellitus (namely, type 1 diabetes), or non insulin-dependent diabetes but there were signs of small vascular disease, Adrenocortical dysfunction is known, malabsorption syndrome is known, and active autoimmune diseases are known.
  17. Other severe acute or chronic medical or psychiatric conditions, or laboratory test abnormalities that may exacerbate the risks associated with participating in or taking test drugs, or that may interfere with the interpretation of test results. These conditions or abnormalities may be determined by the investigator to make the patient unfit to participate in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
DLT | from the start of the medication to the end of the study or 28 days after cessation of medication
  The occurrence of DLT.
AE | from the start of the medication to the end of the study or 28 days after cessation of medication
  The occurrence rate of AE.
ADR | from the start of the medication to the end of the study or 28 days after cessation of medication
  The occurrence rate of adverse drug reactions(ADR).
SAE | from the start of the medication to the end of the study or 28 days after cessation of medication
  The occurrence rate of SAE.
Blood routine | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the laboratory tests.
Urine routine | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the laboratory tests.
Stool routine | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the laboratory tests.
Blood biochemistry | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the laboratory tests.
Coagulation function | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the laboratory tests.
12 lead ecg | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the laboratory tests.
Body temperature | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the vital signs.
Blood pressure | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the vital signs.
Heart rate | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the vital signs.
Breathing | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the vital signs.
General condition | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the physical examination.
Skin | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the physical examination.
Head | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the physical examination.
Eyes | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the physical examination.
Ears | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the physical examination.
Nose | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the physical examination.
Throat | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the physical examination.
Heart | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the physical examination.
Lung | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the physical examination.
Chest | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the physical examination.
Abdomen | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the physical examination.
Limbs | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the physical examination.
Nerves | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the physical examination.
Back/spine | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the physical examination.
Lymph nodes | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the physical examination.

SECONDARY OUTCOMES:
AUCinf | single dose phase:up to 120 hours;multiple dose phase:up to 24 hours
  area under the concentration-time curve from the time of dosing extrapolated to time infinity.
AUC0-24h | single dose phase:up to 24 hours;multiple dose phase:up to 24 hours
  area under the concentration-time curve from the time of dosing extrapolated to the 24h after dosing.
AUC0-72h | single dose phase:up to 72 hours
  area under the concentration-time curve from the time of dosing extrapolated to the 72h after dosing.
AUC0-120h | single dose phase:up to 120 hours
  area under the concentration-time curve from the time of dosing extrapolated to the 120h after dosing.
Peak Plasma Concentration (Cmax) | single dose phase:up to 120 hours;multiple dose phase:up to 24 hours
  The PK parameters of the plasma sample.
CL/F | single dose phase:up to 120 hours;multiple dose phase:up to 24 hours
  The PK parameters of the plasma sample.
Tmax | single dose phase:up to 120 hours;multiple dose phase:up to 24 hours
  The amount of time that a drug is present at the maximum concentration in serum.
Cmin,ss | single dose phase:up to 120 hours;multiple dose phase:up to 24 hours
  The PK parameters of the plasma sample.
Cmax,ss | single dose phase:up to 120 hours;multiple dose phase:up to 24 hours
  The PK parameters of the plasma sample.
Cav,ss | single dose phase:up to 120 hours;multiple dose phase:up to 24 hours
  The PK parameters of the plasma sample.
PTF | single dose phase:up to 120 hours;multiple dose phase:up to 24 hours
  The PK parameters of the plasma sample.
RAUC1 | single dose phase:up to 120 hours;multiple dose phase:up to 24 hours
  The PK parameters of the plasma sample.
RAUC2 | single dose phase:up to 120 hours;multiple dose phase:up to 24 hours
  The PK parameters of the plasma sample.
RCmax | single dose phase:up to 120 hours;multiple dose phase:up to 24 hours
  The PK parameters of the plasma sample.
Kel | single dose phase:up to 120 hours;multiple dose phase:up to 24 hours
  The PK parameters of the plasma sample.
t1/2 | single dose phase:up to 120 hours;multiple dose phase:up to 24 hours
  The PK parameters of the plasma sample.
Vz/F | single dose phase:up to 120 hours;multiple dose phase:up to 24 hours
  The PK parameters of the plasma sample.
AUC_%Extrap | single dose phase:up to 120 hours;multiple dose phase:up to 24 hours
  The PK parameters of the plasma sample.
Ae0-24h | single dose phase:up to 24 hours;multiple dose phase:up to 24 hours
  The PK parameters of the plasma sample.
Fe0-24h | single dose phase:up to 24 hours;multiple dose phase:up to 24 hours
  The PK parameters of the plasma sample.
Ae0-72h | single dose phase:up to 72 hours
  The PK parameters of the plasma sample.
Fe0-72h | single dose phase:up to 72 hours
  The PK parameters of the plasma sample.
Ae0-72h stool | single dose phase:up to 72 hours
  The PK parameters of the plasma sample.
CLr | single dose phase:up to 24 hours;multiple dose phase:up to 24 hours
  The PK parameters of the plasma sample.
Exploring the relative baseline change percentage of biomarkers (soluble VEGFR2). | single dose phase:up to 24 hours;multiple dose phase:up to 24 hours
  The PD parameters of XY0206.
Complete response rate (CRR) | through study completion,such as 30 months.
  Effective parameters of XY0206.
Partial response rate (PRR) | through study completion,such as 30 months.
  Effective parameters of XY0206.
Objective response rate (ORR) | through study completion,such as 30 months.
  Effective parameters of XY0206.
Progression-free survival (PFS) | through study completion,such as 30 months.
  Effective parameters of XY0206.

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, MD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (4):
- China (4):
  - National Cancer Center/Cancer Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Hainan Medical College, Haikou, Hainan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No